CLINICAL TRIAL: NCT02388711
Title: A Randomized Control Trial of the Coordinated-Transitional Care (C-TraC) Intervention for Dementia Patients
Brief Title: A Trial of the C-TraC Intervention for Dementia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2014-1221; 2P50AG033514-06 (NIH); A534255 (Other: UW Madison); SMPH\MEDICINE\GER-AD DEV (Other: UW Madison); Protocol Version 8/21/2018 (Other: UW Madison)
Record Dates: First submitted 2015-02-23; First posted 2015-03-17 (Estimated); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Dementia
Keywords: Dementia; Transitional Care; Caregiver
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care with C-TraC Intervention (Experimental): Patients/caregivers randomized to this group will receive all routine hospital discharge education/materials (same as usual care group), but will also be enrolled in the C-TraC Program. C-TraC is a low-resource, telephone-based, protocol-driven program designed to reduce 30-day rehospitalizations and to improve care transitions during the early post-hospital period.
  Interventions: Other: C-TraC Intervention
- Usual Care (No Intervention): Usual care group patients will receive all routine University of Wisconsin Hospital and Clinics (UWHC) discharge education/materials. This includes pharmacy-led medication teaching, physician discussions and routine nursing education. No post hospital education/contact is performed by these providers. Caregivers are sometimes, but not always, involved. Patients may receive home health services, depending on their physician's discharge plan.

INTERVENTIONS:
Other: C-TraC Intervention — C-TraC utilizes a nurse case manager to coordinate the patient's transitional care through active participation in inpatient multidisciplinary discharge rounds, a single brief protocol-driven inpatient encounter, and 1-4 protocol-driven post-hospital telephone calls with the patient/caregiver using spaced retrieval techniques.
  Arms: Usual Care with C-TraC Intervention

SUMMARY:
The goal of the project is to conduct a prospective, randomized-controlled clinical trial to determine the extent to which the Coordinated-Transitional Care (C-TraC) program impacts transitional care quality, patient cognition/function, caregiver stress and 30-day rehospitalizations in patients with documented diagnoses of dementia discharged from the hospital to the community.

DETAILED DESCRIPTION:
Patients with dementia often experience poor quality transitions from the hospital to the community. In response, the investigators developed and piloted the Coordinated-Transitional Care (C-TraC) program--a low-cost, telephone-based intervention designed to improve care coordination and outcomes in hospitalized patients with dementia or other high-risk conditions discharged to community settings.

A single-blind, prospective, randomized-controlled trial will be used with participants being randomly assigned to receive usual (i.e. standard) care, or usual care plus the C-TraC intervention. Outcomes will be assessed via scheduled phone-calls at 14, 30, and 90 days post-hospitalization. A 45-day phone call will also be conducted to complete a brief satisfaction survey with the caregiver about their post-hospital experience.

ELIGIBILITY:
Patient Inclusion Criteria:

* English-speaking
* Have a working telephone
* Hospitalized on medical inpatient wards at UWHC
* A documented pre-hospitalization diagnosis of dementia.
* Alzheimer's Disease Cooperative Study - Clinical Dementia Rating (ADCS-CDR) score of > 0
* Have a family member/informal caregiver who has regular contact with them in the community setting

Caregiver Inclusion Criteria:

* English-speaking
* Have a working telephone
* Have contact with patient a minimum of once per week

Patient Exclusion Criteria:

* Discharged to institutional settings
* No identified caregiver
* Discharged to hospice
* Followed by complex case management or any form of intensive case management (e.g. transplant, congestive heart failure, dialysis)
* Score moderate-high on modified ASSIST tool for alcohol

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 584 (Actual)
Dates: Start 2015-03; Primary Completion 2019-10-11 (Actual); Study Completion 2019-10-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in rehospitalizations at 14, 30 and 90-days | 14, 30 and 90-days
  The presence of any rehospitalization will be assessed through a combination of 14, 30 and 90 day structured phone calls directly to patients/caregivers, a detailed review of medical records associated with any of these caregiver/patient reported rehospitalizations, and a detailed review of the patient's UWHC medical records after all phone calls are completed.

SECONDARY OUTCOMES:
Increase in patient delirium prevention/resolution | 14, 30 and 90-days
  To assess for delirium, the Family Confusion Assessment Method (FAM-CAM) will be used - an 11-item tool designed to detect delirium from the observations of family caregivers.
Patient functional maintenance/recovery | 14, 30 and 90-days
  To assess function, the investigators will use the Alzheimer's Disease Co-operative Study - Activities of Daily Living Inventory (ADCS-ADL). ADCS-ADL is a 23 item tool which offers detailed descriptions of each functional activity and asks caregivers to describe the patient's observed actions or behaviors.
Patient falls prevention | 14, 30 and 90-days
  Caregivers will be asked to report the presence and dates of any patient falls since discharge.
Decrease caregiver stress | 14, 30 and 90-days
  To measure caregiver stress the 22-item Zarit Caregiver Burden Scale and the 6-item Caregiver Activation Survey (CAS) will be used. The Zarit Caregiver Burden Scale is used as a measure of caregiver psychological stress and the CAS is used as a measure of time spent caregiving.
  The investigators will also assess caregiver stress using the 9-item Patient Health Questionnaire (PHQ-9) and the 3-item Care Transitions Measure (CTM-3). The PHQ-9 is used to establish provisional depressive disorder diagnoses as well as grade the severity of depressive symptoms. The CTM-3 has been modified to be given to caregivers discussing their experience with coordinating their loved ones care after hospital discharge. The statements ask about when the loved one was in the hospital, when they were preparing to leave the hospital and about their medications.

CONTACTS AND LOCATIONS:
Overall Officials: Amy J Kind, MD, PhD, Principal Investigator — University of Wisconsin - Madison, School of Medicine and Public Health, Department of Medicine
Locations (1):
- University of Wisconsin Hospital, Madison, Wisconsin, United States

REFERENCES:
- [Background] Naylor MD, Brooten D, Campbell R, Jacobsen BS, Mezey MD, Pauly MV, Schwartz JS. Comprehensive discharge planning and home follow-up of hospitalized elders: a randomized clinical trial. JAMA. 1999 Feb 17;281(7):613-20. doi: 10.1001/jama.281.7.613. PMID 10029122
- [Background] Naylor MD, Brooten DA, Campbell RL, Maislin G, McCauley KM, Schwartz JS. Transitional care of older adults hospitalized with heart failure: a randomized, controlled trial. J Am Geriatr Soc. 2004 May;52(5):675-84. doi: 10.1111/j.1532-5415.2004.52202.x. PMID 15086645
- [Background] Coleman EA, Parry C, Chalmers S, Min SJ. The care transitions intervention: results of a randomized controlled trial. Arch Intern Med. 2006 Sep 25;166(17):1822-8. doi: 10.1001/archinte.166.17.1822. PMID 17000937
- [Background] Marin DB, Dugue M, Schmeidler J, Santoro J, Neugroschl J, Zaklad G, Brickman A, Schnur E, Hoblyn J, Davis KL. The Caregiver Activity Survey (CAS): longitudinal validation of an instrument that measures time spent caregiving for individuals with Alzheimer's disease. Int J Geriatr Psychiatry. 2000 Aug;15(8):680-6. doi: 10.1002/1099-1166(200008)15:83.0.co;2-7. PMID 10960880
- [Background] Hurd MD, Martorell P, Langa KM. Monetary costs of dementia in the United States. N Engl J Med. 2013 Aug 1;369(5):489-90. doi: 10.1056/NEJMc1305541. No abstract available. PMID 23902508
- [Background] Bourgeois MS, Camp C, Rose M, White B, Malone M, Carr J, Rovine M. A comparison of training strategies to enhance use of external aids by persons with dementia. J Commun Disord. 2003 Sep-Oct;36(5):361-78. doi: 10.1016/s0021-9924(03)00051-0. PMID 12927944
- [Background] Tractenberg RE, Schafer K, Morris JC. Interobserver disagreements on clinical dementia rating assessment: interpretation and implications for training. Alzheimer Dis Assoc Disord. 2001 Jul-Sep;15(3):155-61. doi: 10.1097/00002093-200107000-00007. PMID 11522933